CLINICAL TRIAL: NCT01639989
Title: Pilot Study Which is Aiming at the Feasibility of Performing Doppler Studies of the Spiral Arteries
Brief Title: Doppler Assesment of Blood Flow in the Spiral Arteries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0028-12 HYMC
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Early Pregnancy
Keywords: Doppler, Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study we will try to show that performing Doppler of the Spiral arteries is doable. No outcome will be followed at this stage

DETAILED DESCRIPTION:
This will only be a pilot study to show that we can acurately perform Doppler studies of the spiral arteries

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy 1st trimester

Exclusion Criteria:

* Not willing to participate

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women at 1st trimester
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alon Shrim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel